CLINICAL TRIAL: NCT07218575
Title: A Randomized, Placebo Controlled Double-Blind Trial of Everolimus for Improving Social Abilities in PTEN Germline Mutations
Brief Title: Double-Blind Trial of Everolimus for Improving Social Abilities in PTEN Germline Mutations
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Siddharth Srivastava, Assistant Professor of Neurology, Harvard Medical School, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB-P00049577; 109110 (Other: IND number)
Record Dates: First submitted 2025-10-15; First posted 2025-10-20 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Cowden's Disease; Cowden's Syndrome; Lhermitte-Duclos Disease; Cerebellum Dysplastic Gangliocytoma; Bannayan Zonana Syndrome; Myhre Riley Smith Syndrome; Riley Smith Syndrome; PTEN Hamartoma Tumor Syndrome; Bannayan Riley Ruvalcaba Syndrome
Keywords: PTEN mutation; Autism
MeSH Terms: conditions — Hamartoma Syndrome, Multiple; Autistic Disorder | interventions — Everolimus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Everolimus (Experimental): Everolimus, oral capsules once daily for 12 months; initiated at 2.5mg/day and then increased every 2-3 weeks until a therapeutic blood level is achieved
  Interventions: Drug: Everolimus blinded oral capsules
- Placebo (Placebo Comparator): Placebo matched to everolimus oral capsules once daily for 6 months, Initiated at 1 tablet per day and then increased every 2-3 weeks to maintain blind. Then Everolimus, oral capsules once daily for 6 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Everolimus blinded oral capsules — Oral capsules given once daily for the first 6 months
  Other Names: Afinitor; Zortress
  Arms: Everolimus
Drug: Placebo — Oral capsules given once daily for the first 6 months
  Arms: Placebo

SUMMARY:
The goal of this study is to examine the safety and treatment effects of everolimus in adults and children with PTEN Hamartoma Tumor Syndrome (PHTS) who experience social difficulties. The study will measure if everolimus can safely improve social abilities and functioning in this study population.

PTEN Hamartoma Tumor Syndrome (PHTS) is a genetic condition that results from alteration (germline variant) to the PTEN gene. It is associated with a wide range of symptoms and characteristics, which vary from individual to individual. These include symptoms such as harmatomas (non-cancerous lesions), an increased risk of certain types of cancer, having a larger than average head, and abnormalities in blood vessels. Some people also have neurobehavioral problems including social difficulties. It is estimated approximately 25% (1 in 4) of people with PHTS meet the criteria for an autism diagnosis.

The study lasts for one year. In the first 6 months half of participants will receive everolimus as a once daily oral tablet, and half will receive placebo tablets. For the second 6 months all participants will receive everolimus. Visits to the study clinic are required at the start, month 3, month 6, month 9 and month 12, with phone calls or virtual visits in between. Assessments include questionnaires, blood tests and urine tests, physical and neurological exams, and vital signs.

Everolimus is an existing FDA approved medication used to treat other conditions, including a genetic condition called tuberous sclerosis complex which has some similarities to PHTS, and several types of cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of PTEN Harmartoma Tumor Syndrom (PHTS), confirmed by genetic testing (the testing may be done as part of study screening)
2. Experiences at least moderate levels of social difficulties, based on SRS T score > 60 (measured during screening Have at least a moderate impairment in social abilities, based on SRS score during study screening
3. Fluent in English
4. Females of child-bearing potential must have no plans to become pregnant and be using contraception during the study (if sexually active).
5. Availability of parent, care-giver, partner or other suitable individual who can provide observation reports and provide transportation to attend clinic visits
6. Adequate liver, kidney and bone-marrow function (checked during screening)
7. Medically stable
8. No plans to change school, behavioral therapies, home services or speech therapy during the study period
9. Ability to swallow medicine in pill form

Exclusion Criteria:

1. Ongoing or planned treatment with any medication with known or possible ant-mTOR activity (e.g. sirolimus), or strong inducers or inhibitors of CYP3A, CYP2D6, P450 or PgP (e.g. cyclosporine, ketoconazole, erythromycin, rifampin, phenytoin, phenobarbital) or ACE inhibitors
2. Chronic treatment with systemic corticosteroids or other immunosuppressive treatments (topical or inhaled corticosteroids are allowed).
3. Major surgery or any anti-cancer therapies (including radiotherapy) within 4 weeks of enrollment
4. Neurosurgery within 6 months of enrollment
5. Uncontrolled diabetes defined as HbA1c >8% despite treatment
6. Uncontrolled hyperlipidemia (defined as fasting serum cholesterol > 300 mg/dL OR >7.75 mmol/L AND fasting triglycerides > 2.5 x ULN, assessed during screening)
7. History of Hepatitis B, Hepatitis C or HIV
8. Participation in a clinical trial in the 60 days prior to study entry
9. Known intolerance or hypersensitivity to everolimus or other rapamycin analogs (e.g. sirolimus, temsirolimus)
10. Patients who have a history of another primary malignancy, with the exceptions of non-melanoma skin cancer, and carcinoma in situ of the cervix, uteri, or breast from with the patient has been disease free for > 3 years

Ages: 5 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2030-04 (Estimated); Study Completion 2030-04 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in severity of social skill deficits based on Social Responsiveness Scale (SRS) total score over 6 months. | Baseline, month 1, month 2, month 3, month 4, month 5, month 6
  The SRS is a well-validated, reliable, and widely used measure for identifying and measuring impairments in social processing and associated behaviors. It is completed by an observer who knows the participant well (e.g. parent, care-giver, partner)

SECONDARY OUTCOMES:
Change in overall global clinical assessment of social abilities based on the Clinical Global Impressions (CGI) Improvement scale over 6 months | Month 1, month 2, month 3, month 4, month 5, month 6
  The Clinical Global Impressions (CGI) Improvement rating scale assesses improvement or worsening of symptoms since the start of treatment.
Change from baseline in social skills and processes based on the Stanford Social Dimensions Scale (SSDS) | Baseline, month 1, month 2, month 3, month 4, month 5, month 6
  The Stanford Social Dimensions Scale (SSDS) has been developed to measure an individual's social skills and processes, and is completed by an observer who knows the participant well (e.g. parent, care-giver, partner)
Change from baseline in the Social Communications Sub-scale of the Social Responsiveness Scale (SRS) | Baseline, month 1, month 2, month 3, month 4, month 5, month 6
  The Social Responsiveness Scale (SRS) Social Communication Subscale is part of the SRS questionnaire which is focused on assessment of an individual's ability to communicate and interact with others. It is completed by an observer who knows the participant well (e.g. parent, care-giver, partner)

OTHER OUTCOMES:
Change from baseline in Clinical Global Impression (CGI) Severity Scale | Baseline, month 1, month 2, month 3, month 4, month 5, month 6
  The Clinical Global Impression (CGI) Severity Scale is a rating scale designed to assess severity of symptoms.
Change from baseline in Brief Observation of Social Communication Change (BOSCC) | Baseline, month 6
  The Brief Observation of Social Communication Change (BOSCC) is an instrument that assesses changes in social communication and other autism related social communication behaviors.
Change from baseline in Neurobehavioral Evaluation Tool (NET) - Social Communication and Interaction Subscale | Baseline, month 3, month 6
  The Neurobehavioral Evaluation Tool (NET) is designed to incorporate webcam collected performance measures and informant reported survey responses focusing on autism and other neurobehavioral symptoms. We will evaluate the Social Communication and Interaction Subscale.
Change from baseline in Reading the Mind in the Eyes Test (RMET) | Baseline, month 3, month 6
  The Reading the Mind in the Eyes Test (RMET) is used to evaluate theory of mind, the ability to understand another individual's thoughts.
Change from baseline in Purdue Pegboard Test | Baseline, month 6
  The Purdue Pegboard Test evaluates motor coordination and dexterity.
Change from baseline in Neurobehavioral Evaluation Tool (NET) - Motor subscale | Baseline, month 3, month 6
  The Neurobehavioral Evaluation Tool (NET) is designed to incorporate webcam collected performance measures and informant reported survey responses focusing on autism and other neurobehavioral symptoms. We will evaluate the Motor subscale of this tool.
Change from baseline in Dimensional Assessment of Restricted/Repetitive Behaviors (DARB) | Baseline, month 3, month 6
  The Dimensional Assessment of Repetitive Behaviors (DARB) assess various restricted and repetitive behaviors and interests
Change from baseline in Neurobehavioral Evaluation Tool (NET) - Restricted, Repetitive Behavior subscale | Baseline, month 3, month 6
  The Neurobehavioral Evaluation Tool (NET) is designed to incorporate webcam collected performance measures and informant reported survey responses focusing on autism and other neurobehavioral symptoms. We will evaluate the Restricted, Repetitive Behavior subscale.
Change from baseline in Adult/Child Behavior Checklist (ABCL/CBCL) | Baseline, month 3, month 6
  The Adult/Child Behavior Checklist (ABCL/CBCL) instrument evaluates behavioral and emotional problems in children, adolescents, and adults.
Change from baseline in Neurobehavioral Evaluation Tool (NET) - Disruptive Behaviors subscale. | Baseline, month 3, month 6
  The Neurobehavioral Evaluation Tool is designed to incorporate webcam collected performance measures and informant reported survey responses focusing on autism and other neurobehavioral symptoms. We will evaluate the Disruptive Behaviors subscale.
Change from baseline in Sensory Profile Questionnaire - Short Form | Baseline, month 3, month 6
  The Sensory Profile Questionnaire - Short Form is an assessment of sensory processing features.
Change from baseline in Vineland Adaptive Behavior Scales, 3rd Edition (VABS-3) | Baseline, month 6
  The Vineland Adaptive Behavior Scales, 3rd Edition (VABS-3) characterizes self help skills across a number of different domains.
Change from baseline in Neurobehavioral Evaluation Tool (NET) - Daily Living Skills and Quality of Life Subscales | Baseline, month 3, month 6
  The Neurobehavioral Evaluation Tool (NET) is designed to incorporate webcam collected performance measures and informant reported survey responses focusing on autism and other neurobehavioral symptoms. We will evaluate the Daily Living Skills and Quality of Life subscales.
Change from baseline in Stanford-Binet 5th Edition (SB-5) | Baseline, month 6
  The Stanford-Binet 5th edition (SB-5) is used to characterize various aspects of cognition in children and adults.
Change from baseline in Mullen Scales of Early Learning (MSEL) | Baseline, month 6
  The Mullen Scales of Early Learning (MSEL) is a developmental assessment tool evaluating language, motor, and other abilities.
Change from baseline in Behavior Rating Inventory of Executive Function (BRIEF) | Baseline, month 3, month 6
  The Behavior Rating Inventory of Executive Function (BRIEF) is a tool that evaluates executive functioning in children, adolescents, and adults.
Change from baseline in Neurobehavioral Evaluation Tool (NET) - Executive Functioning subscale | Baseline, month 3, month 6
  The Neurobehavioral Evaluation Tool (NET) is designed to incorporate webcam collected performance measures and informant reported survey responses focusing on autism and other neurobehavioral symptoms. We will evaluate the Executive Functioning subscale.
Change from baseline in the Wide Range Assessment of Memory and Learning-2 (WRAML-2) | Baseline, month 6
  This instrument evaluates memory and cognitive abilities.
Change from baseline in resting state and task-based EEG biomarkers | Baseline, month 6
  Resting state and task-based EEG will also be collected during in person visits to the study sites to examine target engagement of everolimus in the brain.
Change from baseline in eye tracking biomarkers | Baseline, month 3, month 6
  We will assess target engagement in the brain with eye tracking biomarkers
Changes in total/phosphorylated PTEN-associated protein levels | Screening visit, month 6
  We will examine if PTEN-associated molecules (mTOR, MAPK, PI3K/AKT) are affected by everolimus, and assess changes with treatment in total/phosphorylated protein levels from peripheral blood mononuclear cells.